CLINICAL TRIAL: NCT03347292
Title: A Multicenter, Non-randomized, Open-label Dose Escalation Phase Ib Study of Regorafenib in Combination With Pembrolizumab in Patients With Advanced Hepatocellular Carcinoma (HCC) With no Prior Systemic Therapy
Brief Title: Regorafenib Plus Pembrolizumab in First Line Systemic Treatment of HCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19497; KN-743 (Other: Merck Sharp & Dohme); 2017-003202-40 (EudraCT Number)
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Liver cell carcinoma; Liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — regorafenib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): The regorafenib starting dose will be 120 mg q.d.(once daily) 3 weeks on / 1 week off in combination with the recommended dose of pembrolizumab (200 mg Q3W). Pembrolizumab dose will not be escalated or de-escalated.
  Interventions: Drug: Regorafenib(Stivarga, BAY73-4506); Drug: Pembrolizumab
- Dose expansion (Experimental): Dose expansion cohorts will continue to be expanded until the sample size of 30-35 patients per cohort is reached.
  Interventions: Drug: Regorafenib(Stivarga, BAY73-4506); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Regorafenib(Stivarga, BAY73-4506) — Regorafenib 80mg/120mg/160mg q.d., 3 weeks on / 1 week off + pembrolizumab 200mg i.v. every 3 weeks
Drug: Pembrolizumab — 200 mg i.v.(Intravenous(ly)) every 3 weeks (Q3W). This dose will not be escalated or deescalated and the dosing schedule will not be changed

SUMMARY:
This study will determine if the combination of regorafenib and pembrolizumab is safe and tolerated in patients with advanced liver cancer. In addition, the study will explore the anti-tumor activity of this combination as well as potentially identifying blood and tissue biomarkers associated with disease activity, status or response. The study will also investigate how the drugs behave in your body

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age on day of signing informed consent.
* Histological or cytological confirmation of HCC (hepatocellular carcinoma) or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases (AASLD) criteria in patients with a confirmed diagnosis of cirrhosis.
* Barcelona Clinic Liver Cancer (BCLC) stage B or C that cannot benefit from treatments of established efficacy such as resection, local ablation, chemoembolization.
* Liver function status Child-Pugh (CP) Class A. CP status should be calculated based on clinical findings and laboratory results during the screening period.
* Any local or loco-regional therapy of intrahepatic tumor lesions (e.g. surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed ≥ 4 weeks before first dose of study medication. Note: patients who received sole intrahepatic intra-arterial chemotherapy, without lipiodol or embolizing agents are not eligible.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* At least one uni-dimensional measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST (RECIST version 1.1) and no older than 28 days before start of the study treatment. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if there has been demonstrated progression in the lesion.
* Life expectancy of at least 3 months.
* Adequate bone marrow and organ function as assessed by the laboratory tests performed within 7 days before of treatment initiation.
* For patients recruited in the expansion cohort only, provision of archival (block) or fresh tumor tissue samples at baseline is mandatory. If archival tumor tissue is not available, patients should be willing to undergo a biopsy for provision of fresh tumor samples

Exclusion Criteria:

* Prior systemic therapy for HCC; prior exposure to regorafenib.
* Previous treatment with a programmed death 1 (PD1), programmed death-ligand (PD-L1), or cytotoxicT-lymphocyte-associated protein 4 (CTLA-4) inhibitors, or any form of immunotherapy for HCC.
* Previous treatment with live vaccine within 30 days of planned start of study drugs (seasonal flu vaccines that do not contain a live virus are permitted).
* Active autoimmune disease (active defined as having autoimmune disease related symptoms and detectable autoantibodies) that has required systemic treatment in the past 2 years (i.e., with use of diseasemodifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drugs. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
* Known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies).
* Dual active HBV infection (HBsAg (+) and /or detectable HBV DNA) and HCV infection (anti-HCV Ab(+) and detectable HCV RNA) at study entry.
* Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE Grade 2 dyspnea).
* Known history of metastatic brain or meningeal tumors.
* Significant acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease,malabsorption, or CTCAE Grade ≥ 2 diarrhea of any etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse event(TEAEs) | Up to 30 days after last dose of study drug
  The incidence of treatment-emergent adverse events and treatment-emergent drug-related adverse events summarized in frequency tables using worst CTCAE v4.03 grade.
Severity of TEAEs | Up to 30 days after last dose of study drug
Dose Limiting Toxicities(DLTs) | Up to 42 days after first treatment administration

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) | After approximately 18 months
  The MTD is defined as the highest dose that can be given so that toxicity probability is below the target toxicity PT =35%.
Progression-free survival (PFS) | After approximately 36 months
Time to progression (TTP) | After approximately 36 months
Overall survival (OS) | After approximately 36 months
Overall response rate (ORR) | After approximately 36 months
Disease control rate (DCR) | After approximately 36 months
Duration of response (DOR) | After approximately 36 months
Duration of stable disease | After approximately 36 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - USC Norris Hospital and Clinics, Los Angeles, California
  - University of Florida Health Sciences Center, Gainesville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Mount Sinai Medical Center, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
- Germany (2):
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.